CLINICAL TRIAL: NCT03902353
Title: Screening of Pulmonary Veino Occlusive Disease in Heterozygous EIF2AK4 Mutation Carriers
Acronym: DELPHI-4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K180501J
Record Dates: First submitted 2019-03-14; First posted 2019-04-04 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2019-07

CONDITIONS: Mutation; Genetic Syndrome
Keywords: Pulmonary veino occlusive disease, pulmonary hypertension
MeSH Terms: conditions — Genetic Diseases, Inborn; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults without diagnosis of PH (Other): Adults without diagnosis of PH carrying an heterozygous EIF2AK4
  Interventions: Other: Screening of adult without diagnosis of PH carrying an heterozygous EIF2AK4 mutation.

INTERVENTIONS:
Other: Screening of adult without diagnosis of PH carrying an heterozygous EIF2AK4 mutation. — will be performed : a clinical evaluation (dyspnea assessed by New York Heart Association functional class (I-IV), signs of right heart failure), a 6min walk test, a Computerized Tomography scan of the chest, an electrocardiogram, an echocardiography (measurement of the velocity of tricuspid regurgitation, measurement of Tricuspid Annular Plane Systolic Excursion (TAPSE) and Tei index, pericardial effusion, dilatation and hypertrophy of the right ventricle), an abdomina ulstrasound, a stress Test (ventilation oxygen peak and ventilation oxygen specific, minute ventilation, dead-space ventilation / dead space, ventilatory reserve, alveolar-arterial gradient, pulse oxygen, PaO2), a lung function tests and measurement of Diffusing capacity or transfer factor of the Lung for Carbon mOnoxide (DLCO) and Nitric Oxide (DLNO), and a blood sample.

SUMMARY:
Pulmonary Veino Occlusive Disease (PVOD) is a rare form of pulmonary arterial hypertension, characterised by a poor prognosis. Recent studies demonstrated that heritable form of pulmonary veino occlusive diseaseis due to bi-allelic mutations in EIF2AK4 gene. heritable pulmonary veino occlusive disease is an autosomal recessive disease. In the french referal center of severe PH, ulmonary veino occlusive disease patients carriers of bi-allelic mutations in EIF2AK4 gene were identified. Genetic counselling in these families allowed to identified herozygous carriers of a single mutation in EIF2AK4 gene. However, to date, nothing is known about the risk of these persons of developping pulmonary diseases. It appears essential to determine the clinical, functional, echocardiographic and radiologics characteristics of these persons, and their risk of developping Pulmonary veino occlusive disease

DETAILED DESCRIPTION:
the investigators will evaluate the subjects at inclusion after informed by a clinical evaluation (dyspnea assessed by New York Heart Association functional class (I-IV), signs of right heart failure), a 6min walk test, a Computerized Tomography scan of the chest, an electrocardiogram, an echocardiography , an abdomina ulstrasound, a Cardiopulmonary exercise testing, a lung function tests , arterial blood gases.

At one and two years, a phone call will be made to to participants evaluate dyspnea and intercurrent events in all subjects. In the presence of pulmonary veino occlusive diseaseis symptoms, a new evaluation will be proposed in order to confirm of not pulmonary veino occlusive diseaseis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult (age ≥18 years of age at the date of inclusion),
* With an identification of the presence of a mutation of the EIF2AK4 gene in the heterozygous state,
* Having given free and informed consent.

Exclusion Criteria:

* Minor (age <18 years),
* Patient with known Pulmonary veino occlusive disease or Pulmonary arterial hypertension
* Woman having started a pregnancy or breastfeeding
* protected adult persons,
* Persons deprived of their liberty,
* People in emergency,
* Those who refused or were unable to give informed consent,
* Contraindication to the exercise test (acute coronary syndrome, syncope, tight stenotic valve disease ...) See the list of relative and absolute contraindications to the exercise test (chapter 6.2).
* No affiliation to a social security scheme (beneficiary or beneficiary).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of characteristics of asymptomatic heterozyous EIF2AK4 mutation carriers and monitor these subjects' clinical, functional, biological, echocardiographic | 1 year
  frequency of abnormalities observed

SECONDARY OUTCOMES:
predictive factors of the occurrence of PVOD follow prospectively a cohort of asymptomatic heterozyous EIF2AK4 mutation carriers to determine predictive factors of the occurrence of VOD | 1 year
  number of heterozygous EIF2AK4 mutation carriers who will develop Pulmonary Veno-Occlusive Disease

CONTACTS AND LOCATIONS:
Overall Officials: MONTANI David, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- David MONTANI, Le Kremlin-Bicêtre, Krémlin Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lechartier B, Girerd B, Eyries M, Beurnier A, Humbert M, Montani D. Screening for pulmonary veno-occlusive disease in heterozygous EIF2AK4 variant carriers. Eur Respir J. 2022 Aug 18;60(2):2200760. doi: 10.1183/13993003.00760-2022. Print 2022 Aug. No abstract available. PMID 35710265